CLINICAL TRIAL: NCT04698421
Title: Prospective Collection of Biological Samples from Patients with Rare Neurological Diseases
Brief Title: Collection of Biological Samples from Patients with Rare Neurological Diseases
Acronym: EXPLAINEUR
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/20/0150
Record Dates: First submitted 2020-12-23; First posted 2021-01-06 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Nervous System Diseases
Keywords: autoimmune encephalitis; paraneoplastic neurological syndrome; myasthenia; paraneoplastic cerebellar degeneration; rare neuropathologies with known/suspected autoimmune origin
MeSH Terms: conditions — Nervous System Diseases; Autoimmune Diseases of the Nervous System; Paraneoplastic Cerebellar Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- patients with rare autoimmune neurological diseases
  Interventions: Biological: Blood collection on admission and longitudinally

INTERVENTIONS:
Biological: Blood collection on admission and longitudinally — Biological samples will be collected in the normal diagnosis and follow-up process. Only blood will be taken in larger quantity (8 tubes of 7mL).

SUMMARY:
The aim of this project is to improve biological collections of patients presenting rare neurological disorders with known or suspected autoimmune origin. This collection will provide appropriate biological samples to identify new biomarkers and to be accessible to the medical, scientific and industrial communities for the identification of new therapeutic strategies.

DETAILED DESCRIPTION:
Neuroimmunology is a rapidly expanding field since major advances have been made in basic immunology and numerous new clinical entities have been identified in the last 10 years. Even if these discoveries have led to major advances in patient's management and treatment, a lot of work needs to be done to improve the diagnosis and prognostic biomarkers. It is widely known that the immune system is implicated in a variety of neurological disorders such as infections, encephalitis or multiple sclerosis. Numerous neurological disorders affecting the central and peripheral nervous system can be attributed to the immune system and need to be recognized as some of them can be cured by appropriate immunotherapy. These neurological disorders include autoimmune encephalitis and paraneoplastic neurological syndromes but also myasthenia, chronic demyelinating inflammatory polyneuropathy and other neuromuscular pathologies.

These neurological disorders are characterized by the presence of autoantibodies in the patient's sera or cerebral spinal fluid (CSF). These autoantibodies are generally highly specific and necessary to make the diagnosis. However, in some cases, despite strong clinical arguments for a neuroimmunological disorder, we do not identify autoantibodies, leading to inappropriate treatment and a blind follow-up considering the risk of recurrence or of associated tumor. Furthermore, even if the specific role of some autoantibodies or of immune T cells in some of these pathologies are suspected or already documented, for most of them the exact mechanism is still unknown. We need to explore the sera and CSF of these patients to identify new diagnosis and prognosis biomarker. Moreover, the availability of immune cells isolated from these patients will help us to decipher the pathophysiological mechanisms to create new therapeutic strategies. For this, animal models are already available in Centre Physiopathology Toulouse and in the French reference center in Lyon. As genetic susceptibilities may underlie, at least in part, the variability of the clinical manifestations and of the response to treatment, DNA from patients will be collected and immune genes sequencing will be compared to other control groups, included international database.

ELIGIBILITY:
Inclusion Criteria:

* all patients with neurological disorders, with known or probable autoimmune involvement. This includes adults and children and peripheral and/or central nervous system symptoms.
* Social coverage up to date.

Exclusion Criteria:

* Patients with neurological damage from which the autoimmune character can be excluded.
* Known anemia and hemoglobin <10 g / dl
* Patients under protective supervision (guardianship, curators)
* Pregnant or breastfeeding woman

Ages: 6 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients followed at the Toulouse University Hospital and presenting rare neurological disorders with known or suspected autoimmune origin
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-10-12 (Actual); Primary Completion 2030-01-01 (Estimated); Study Completion 2030-09-03 (Estimated)

PRIMARY OUTCOMES:
Building a collection of biological samples and clinical-biological data from patients with rare autoimmune neurological diseases | Day 0 and through study completion, an average of 1 year
  Blood sampling

SECONDARY OUTCOMES:
Identification of new autoantibodies. | Day 0 and through study completion, an average of 1 year
  ELISA
Identification of biomarkers regarding the severity (such as cytokines, axonal damages...) in order to help the therapeutic decisions. | Day 0 and through study completion, an average of 1 year
  Analysis of the phenotypic profiling of blood immune cells by multicolor fluorescence-activated cell sorter (FACS) analysis and of the transcriptomic profiling of blood immune cells by RNA sequencing
Exploration of the pathophysiological mechanisms of rare autoimmune neurological pathologies. | Day 0 and through study completion, an average of 1 year
  Knock-out or knock-in animal models for one specific protein will be used to determine in vivo if the pathophysiological mechanisms of rare autoimmune neurological disorder can be induced by the abnormal expression of this protein.

CONTACTS AND LOCATIONS:
Overall Officials: Chloé Bost, PharmD, PhD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Purpan University Hospital, Toulouse, France

IPD SHARING:
Plan to Share IPD: No